CLINICAL TRIAL: NCT01228968
Title: Toward an Automated Method of Abdominal Fat Segmentation of MR Images
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: MRImethods060229
Record Dates: First submitted 2010-10-25; First posted 2010-10-27 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Obesity
Keywords: obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Volunteers: Volunteers will have a range of body mass index from 19 - 45 kilogram per square meter. In order to fit in the magnetic resonance scanner subjects must weigh less than 300 pounds.

SUMMARY:
Subjects will undergo a brief magnetic resonance (MRI) scan. The resulting images will be used to compare two abdominal fat segmentation techniques. The first technique is already validated and in use. The second technique was recently developed and has not been validated. The hypothesis is that the second technique will be the faster and more reliable of the two.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory
* cognitively sound

Exclusion Criteria:

* body mass index less than 18 or greater than 45 kilograms per square meter

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will have a wide range of body mass index and other physical characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: we recruited subjects currently enrolled in related studies.
Period: Overall Study
Arm/Group | Volunteers
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Volunteers
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Secondary Outcome: Subcutaneous Fat Volume With Automated Analysis
Description: This is the volume of Abdominal Subcutaneous Fat in cubic centimeters as determined with new automated anatomical segmentation software.
Time Frame: five minutes
Measure: Mean (Standard Deviation); unit: cubic centimeters
Arm/Group | Volunteers
Number analyzed (Participants) | 9
cubic centimeters | 2506 (887)

2. Primary Outcome: Visceral Fat Volume With Automated Analysis
Description: This is the measurement of Abdominal Visceral Fat in cubic centimeters as determined with a new automated segmentation program.
Time Frame: five minutes
Measure: Mean (Standard Deviation); unit: cubic centimeters
Arm/Group | Volunteers
Number analyzed (Participants) | 9
cubic centimeters | 994 (618)

3. Primary Outcome: Visceral Fat Volume With Manual Segmentation
Description: This is the measure of visceral fat found with our older manual segmentation method
Time Frame: five minutes
Measure: Mean (Standard Deviation); unit: cm3
Arm/Group | Volunteers
Number analyzed (Participants) | 9
cm3 | 1175 (636)

4. Secondary Outcome: Subcutaneous Fat Volume With Manual Segmentation
Description: This is the volume of Abdominal Subcutaneous Fat in cubic centimeters as determined with the older manual segmentation technique.
Time Frame: five minutes
Measure: Mean (Standard Deviation); unit: cubic centimeters
Arm/Group | Volunteers
Number analyzed (Participants) | 9
cubic centimeters | 2910 (964)

ADVERSE EVENTS:
Arm/Group | Volunteers
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No